CLINICAL TRIAL: NCT06442436
Title: A Study to Evaluate the Pharmacokinetics of Nemtabrutinib in Participants With Moderate Hepatic Impairment
Brief Title: A Study of Nemtabrutinib in Participants With Moderate Hepatic Impairment (MK-1026-015)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1026-015; MK-1026-015 (Other: MSD)
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Hepatic Impairment (HI)
MeSH Terms: interventions — ARQ531

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Panel A (Experimental): Participants with moderate hepatic impairment will receive a single oral dose of 25 mg nemtabrutinib on Day 1.
  Interventions: Drug: Nemtabrutinib
- Panel B (Experimental): Healthy control participants will receive a single oral dose of 25 mg nemtabrutinib on Day 1.
  Interventions: Drug: Nemtabrutinib

INTERVENTIONS:
Drug: Nemtabrutinib — 25 mg nemtabrutinib (1 x 5 mg and 1 x 20 mg tablets) administered orally as a single dose.
  Other Names: MK-1026; ARQ 531

SUMMARY:
The purpose of this study is to compare the plasma pharmacokinetics (PK) of nemtabrutinib (MK-1026) following a single oral dose of nemtabrutinib in participants with moderate hepatic impairment to that of healthy matched control participants and to evaluate the safety and tolerability of nemtabrutinib.

ELIGIBILITY:
Inclusion Criteria:

* Has a body mass index (BMI) between 18.0 and 40.0 kg/m2, inclusive.
* Is assigned male or female sex at birth. Participants assigned female sex at birth must not be pregnant or breast feeding and must be of nonchild bearing potential.
* Who agrees to use contraception.
* Has provided documented informed consent for the study.
* Has a diagnosis of chronic (>6 months), stable (no acute episodes of illness within the previous 2 months due to deterioration in hepatic function) hepatic impairment with features of cirrhosis due to any etiology (moderate HI only).
* Has moderate hepatic impairment (class B) by the Child-Pugh classification system AND/OR the participant has moderate impairment by the National Cancer Institution Organ Dysfunction Working Group (NCI-ODWG) classification system (moderate HI only).
* Is in general good health (except for Moderate HI).

Exclusion Criteria:

* Has a clinically significant condition that may affect absorption of the study drug in the opinion of the investigator, including gastric restrictions and bariatric surgery (eg, gastric bypass).
* Is mentally or legally incapacitated, has significant emotional problems at the time of prestudy (screening) visit or expected during the conduct of the study or has a history of clinically significant psychiatric disorder of the last 5 years.
* Has a history of cancer (malignancy).
* Has a history of significant multiple and/or severe allergies (eg, food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability (systemic allergic reaction) to prescription or nonprescription drugs or food.
* Had a major surgery and/or donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the prestudy.
* Has received any vaccine starting from 14 days prior to study or is scheduled to receive any vaccine through 30 days following study intervention.
* Was dosed in another investigational study within 4 weeks (or 5 half-lives, whichever is greater) prior to check-in (Day -1).
* Is under the age of consent.
* Is heavy smoker or heavy user of nicotine-containing products (>20 cigarettes or equivalent/day).
* Is regular user of cannabis or any illicit drugs or has a history of drug (including alcohol) abuse within approximately 3 months.
* Consumes greater than 3 servings of alcoholic beverages per day.
* Consumes excessive amounts, defined as greater than 6 servings of coffee, tea, cola, (1 serving is approximately equivalent to 120 mg of caffeine) energy drinks, or other caffeinated beverages per day.
* Is unwilling to comply with the study restrictions.
* Has a history or illness that in the opinion of the investigator, might confound the results of the study or poses an additional risk to the participant by their participation in the study (moderate HI only).
* Has a history of recent variceal bleeds (for moderate HI only).
* Has evidence of hepatorenal syndrome (for moderate HI only).
* Has fluctuating or rapidly deteriorating hepatic function within the prestudy period, in the opinion of the investigator (for moderate HI only).
* Is not in sufficient health, with regard to stability of HI, to undergo participation in the study with anticipated survival of <3 months, in keeping with a Model for End-Stage Liver Disease (MELD) score of ≥25 (for moderate HI only).
* Has a history of liver or other solid organ transplantation (for moderate HI only).
* Has an active infection requiring systemic therapy (for moderate HI only).
* Who requires paracentesis more often than 2 times per month (for moderate HI only).
* Has a transjugular intrahepatic portosystemic shunt and/or has undergone portacaval shunting (for moderate HI only).
* Has encephalopathy Grade 3 or worse within 28 days before administration of study intervention (for moderate HI only).
* Has received antiviral and/or immune modulating therapy for hepatitis B virus (HBV) or hepatitis C virus (HCV) within 90 days prior to study start (for moderate HI only).
* Is positive for human immunodeficiency virus (HIV)-1 or HIV-2 or using HIV protease inhibitors (for moderate HI only).
* Is positive for HBV (for moderate HI only).
* Is positive for HCV (for moderate HI only).
* Is taking medications to treat chronic medical conditions and has not been on a stable regimen for at least 1 month and/or is unable to withhold the use of the medication(s) for the prohibited period of time in study (for moderate HI only).
* Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological (history of a bleeding disorder, abnormal bleeding or a hereditary or acquired coagulation or platelet disorder), hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke, intracranial hemorrhage, and chronic seizures) abnormalities or diseases (for healthy control participants only).
* Has positive test(s) for hepatitis B surface antigen (HBsAg), hepatitis C antibodies, or HIV at the prestudy (screening) visit (for healthy control participants only).
* Is unable to refrain from or anticipates the use of any medication, including prescription and nonprescription drugs or herbal remedies (for healthy control participants only).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2026-09-14 (Estimated); Study Completion 2026-09-14 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve from Dosing to Infinity (AUC0-inf) of Nemtabrutinib in Plasma | Predose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 192, 240, and 336 hours postdose
  The AUC0-inf of nemtabrutinib in plasma will be determined in each arm.
Maximum Concentration (Cmax) of Nemtabrutinib in Plasma | Predose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 192, 240, and 336 hours postdose
  The Cmax of nemtabrutinib in plasma will be determined in each arm.

SECONDARY OUTCOMES:
Area Under the Curve from Dosing to last (AUC0-last) of Nemtabrutinib in Plasma | Predose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 192, 240, and 336 hours postdose
  The AUC0-last of nemtabrutinib in plasma will be determined in each arm.
Concentration 24 (C24) Hours Postdose of Nemtabrutinib in Plasma | 24 hours postdose
  The C24 of nemtabrutinib in plasma will be determined in each arm.
Time to Maximum Concentration (Tmax) of Nemtabrutinib in Plasma | Predose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 192, 240, and 336 hours postdose
  The Tmax of nemtabrutinib in plasma will be determined in each arm.
Apparent Terminal Half-life (t1/2) of Nemtabrutinib in Plasma | Predose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 192, 240, and 336 hours postdose
  The t½ of nemtabrutinib in plasma will be determined in each arm.
Apparent Total Clearance (CL/F) of Nemtabrutinib in Plasma | Predose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 192, 240, and 336 hours postdose
  The CL/F of nemtabrutinib in plasma will be determined in each arm.
Apparent Volume of Distribution During Terminal Phase (Vz/F) of Nemtabrutinib in Plasma | Predose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 192, 240, and 336 hours postdose
  The Vz/F of nemtabrutinib in plasma will be determined in each arm.
Number of Participants who Experience One or More Adverse Events (AEs) | Up to ~15 days
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants experiencing AEs will be reported.
Number of Participants Who Discontinue From the Study Due to an Adverse Event (AE) | Up to ~15 days
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants discontinuing study treatment due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (3):
- United States (3):
  - Clinical Pharmacology of Miami ( Site 0003), Miami, Florida
  - Orlando Clinical Research Center ( Site 0001), Orlando, Florida
  - Texas Liver Institute ( Site 0002), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com